CLINICAL TRIAL: NCT01154166
Title: A Phase III, Randomised, Double-blind, Placebo-controlled, Parallel Group Study of Six Months Treatment With Ropinirole PR as Adjunctive Therapy in Patients With Parkinson's Disease Who Are Not Optimally Controlled on L-Dopa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111528
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2012-08-07 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ReQuip PR (Experimental): Ropinirole PR tablets of 2.0 mg, 4.0mg and 8.0 mg
  Interventions: Drug: ReQuip PR
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ReQuip PR — If subjects are still eligible at the end of the placebo run-in period they will be randomized (1:1) to receive once daily doses of ropinirole PR or identical appearing placebo tablets. Dosing will start at 2 mg ropinirole PR, or placebo equivalent. During the 24 week treatment phase, the subjects dose will be adjusted according to the recommended schedule to achieve symptomatic control. All subjects must be titrated to a minimum dose of 6 mg/day.
  Arms: ReQuip PR
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a phase III, multicenter, randomized, double-blind, parallel group, placebo-controlled study to compare the efficacy of 6-months therapy of ropinirole Prolonged Release (PR) with that of placebo as adjunctive therapy to L-dopa in Parkinson's disease patients not optimally controlled on L-dopa. This study will be conducted in China. Subjects will have total 14 visits over the 26 week duration of the study.

Following screening, eligible subjects will receive study medication during the fourteen day placebo run-in period which they will be instructed to take in addition to their background L-dopa. If subjects are still eligible at the end of the placebo run-in period they will be randomized (1:1) to receive once daily doses of ropinirole PR or identical appearing placebo tablets. Dosing will start at 2 mg ropinirole PR, or placebo equivalent. During the 24 week treatment phase, the subjects dose will be adjusted according to the recommended schedule to achieve symptomatic control. All subjects must be titrated to a minimum dose of 6 mg/day. If sufficient symptomatic control is not achieved or maintained at a dose of 6mg/day of ropinirole PR, the daily dose should be increased by 2mg at weekly or longer intervals up to a dose of 8mg/day.If sufficient symptomatic control is still not achieved or maintained at a dose of 8mg/day of ropinirole PR, the daily dose should be increased by 4mg at two weekly or longer intervals. Further dose titration should not be conducted within the final 8 weeks of the treatment phase. The maximum recommended daily dose is 24mg.

The planned reduction in L-dopa dose will begin once subjects are titrated to Dose Level 4 or Dose Level 5 of study medication. For each increase in study medication, there will be a corresponding decrease in L-dopa. If loss of symptom control occurs with the reduction in the background L-dopa dose, the dose of study medication should be increased to the next higher dose level with no adjustment in the dose of L-dopa. If loss of symptom control persists, subjects should be titrated up an additional dose level. Subjects who do not experience an improvement in symptoms following upward titration by 2 dose levels of study medication, should be "rescued" with L-dopa.

Subjects will be dispensed down-titration medication at the study completion/early withdrawal visit if the patient did not enter extension study and should be scheduled to return for a follow up visit 4 to 14 days after the last dose of study medication. The extension study aim to evaluate the safety profile of ReQuip PR during long-term treatment in subjects with advanced parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Men or non-pregnant/non-breast-feeding women of at least 30 years of age at screening.Women of child-bearing potential must be practicing a clinically accepted method of contraception (such as oral contraception, surgical sterilization, intrauterine device [IUD], or diaphragm IN ADDITION to spermicidal foam and condom on male partner, or systemic contraception [i.e. Norplant System]), during the study and for at least one month prior to randomisation and one month following completion of the study.
* Diagnosis of idiopathic Parkinson's Disease (according to modified Hoehn & Yahr criteria Stages II-IV) and demonstrating lack of control with L-dopa therapy (e.g. end of dose akinesia, simple on/off fluctuations)
* Subjects receiving a stable dose of L-dopa for at least four weeks prior to screening.
* Provide written informed consent for this study
* A minimum of 3 hours awake time"off " for each diary day recorded during the Placebo Run-In Period.
* Be willing and able to comply with study procedures, including diary card completion and follow-up clinic visits.

Exclusion Criteria:

* Late stage advanced subjects demonstrating incapacitating peak dose or biphasic dyskinesia on their stable dose of L-dopa.
* Presence, or history within the previous 3 months, of significant and/or uncontrolled psychiatric, hematological, renal, hepatic, endocrinological, neurological (other than Parkinson.s Disease), or cardiovascular disease or active malignancy (other than basal cell cancer);
* Any abnormality, at Screening, that the investigator deems to be clinically relevant on history, physical examination and in diagnostic laboratory tests including ECG;
* Unstable liver disease, cirrhosis, known biliary abnormalities(except Gilbert's syndrome or asymptomatic gallstones) or AST or ALT>2xULN or alk phos and bilirubin>1.5 xULN
* Recent history of severe dizziness or fainting due to postural hypotension on standing.
* Clinical dementia that in the judgment of the investigator would preclude assessment of the subject.
* Recent history or current evidence of drug abuse or alcoholism.
* Consumption of any dopamine agonist within four weeks of the screening visit.
* Definite or suspected personal or family history of clinically significant adverse reactions or hypersensitivity to ropinirole (or to drugs with a similar chemical structure) that would preclude long-term dosing with ropinirole PR.
* Withdrawal, introduction, or change in dose of hormone replacement therapy and/or any drug known to substantially inhibit CYP1A2 (e.g. ciprofloxacine, fluvoxamine, cimetidine, ethinyloestradiol) or induce CYP1A2 (e.g. tobacco, omeprazole) within 7 days prior to enrolment. Subjects already on chronic therapy with any of these agents may be enrolled but must remain on stable doses of the agent from 7 days prior to enrolment through the end of the Treatment Period.
* Use of an investigational drug within 30 days or 5 half-lives (which ever is longer).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2010-02-15; Primary Completion 2011-09-01 (Actual); Study Completion 2011-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- China (10):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Suzhou, Jiangsu
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Kunming, Yunnan
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 347 participants were randomized; however, 2 participants were not dosed after randomization and were excluded from the Safety Population. An additional participant had no post-baseline assessment available and was thus excluded from the Intent-to-Treat Population. Thus, only 344 of the 347 randomized participants "started" the study.
Pre-assignment Details: After the 14-day Run-in Phase with placebo, eligible participants (par.) entered the 24-week Treatment Phase (TP) and were randomized 1:1 to ropinirole PR or placebo. After the TP, all par. were down-titrated for 7 days. Those who did not enter the extension study returned for a follow-up visit 4-14 days after the last dose of medication.
Groups:
- Placebo: Participants received placebo tablets identical to ropinirole prolonged release (Ro-PR) tablets once daily (OD) in the 24-week Treatment Phase (TP). The L-dopa dose was reduced after a dose of 8 milligrams (mg) or 12 mg of study medication had been achieved. If a loss of symptom control occurred and persisted after study medication had been up-titrated once, participants were to be "rescued" with open-label L-dopa, which was not to exceed the dose being taken at baseline. After the 24-week TP, all participants were down-titrated over a 7-day period. Those participants who did not enter the extension study returned for a follow-up visit 4 to 14 days after the last dose of medication.
- Ropinirole PR: Participants initially received Ro-PR 2 mg tablets OD in the 24-week TP. The Ro-PR dose was up-titrated weekly by 2 mg for the first 3 weeks of treatment. Later, the daily dose was increased by 4 mg every 2 weeks, up to a maximum dose of 24 mg per day. The L-dopa dose was reduced after a dose of 8 mg or 12 mg of study medication had been achieved. Participants who did not experience symptom improvement after up-titration of Ro-PR by 2 dose levels were allowed to take L-dopa (maximum up to their baseline dose). After the 24-week TP, all participants were down-titrated over a 7-day period. Those participants who did not enter the extension study returned for a follow-up visit 4 to 14 days after the last dose of Ro-PR.
Period: Overall Study
Arm/Group | Placebo | Ropinirole PR
Started | 169 | 175
Completed | 135 | 163
Not Completed | 34 | 12
Not completed — Adverse Event | 14 | 9
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 4 | 1
Not completed — Withdrawal by Subject | 10 | 1
Not completed — Lack of Efficacy | 3 | 0
Not completed — Disease Progression | 1 | 0
Not completed — Poor Compliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ropinirole PR | Total
Number analyzed (Participants) | 169 | 175 | 344
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline data were collected in members of the Intent-to-Treat (ITT) Population, comprised of all randomized participants who received at least one dose of study medication and for whom at least one post-baseline efficacy assessment was available.
  Years | 63.6 (10.50) | 64.1 (8.99) | 63.9 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline data were collected in members of the Intent-to-Treat (ITT) Population, comprised of all randomized participants who received at least one dose of study medication and for whom at least one post-baseline efficacy assessment was available.
  Participants
    Female | 65 | 59 | 124
    Male | 104 | 116 | 220
Race/Ethnicity, Customized [Number; unit: participants] — Baseline data were collected in members of the Intent-to-Treat (ITT) Population, comprised of all randomized participants who received at least one dose of study medication and for whom at least one post-baseline efficacy assessment was available.
  participants
    Oriental | 169 | 175 | 344

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Total Awake Time Spent "Off" at Week 24 Using Last Observation Carried Forward (LOCF)
Description: The "off" state is defined as the state in which Parkinson's Disease (PD) symptoms (lack of mobility, tremor, or rigidity) are not adequately controlled by the drug. Participants were asked to record the duration of their "off " periods in 24-hour diary cards prior to each visit on two days of each relevant week. The total number of awake hours spent "off" per 24-hour period was the sum of the hours recorded on the two 24-hour diary cards. Change from Baseline is calculated as the value at Week 24 minus the Baseline value.
Time Frame: Baseline and Week 24 (Visit 13)
Population: Intent-to-treat (ITT) Population: all randomized participants who received at least one dose of study medication and for whom at least one post-baseline efficacy assessment was available. In the LOCF dataset, the last available on-therapy observation for a participant is used to estimate missing data points.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | Ropinirole PR
Number analyzed (Participants) | 169 | 175
hours | -0.4 (2.47) | -2.1 (2.58)
Statistical Analysis 1: Comparison: Placebo vs Ropinirole PR; Test type: Superiority or Other; p < 0.001, ANCOVA; Adjusted mean for treatment difference = -1.76, 95% CI 2-sided [-2.27 to -1.26] — The estimated value indicates the treatment difference for the adjusted mean for Ropinirole PR and placebo

2. Secondary Outcome: Mean Change From Baseline (BL) in the Unified Parkinson Disease Rating Scale (UPDRS) Total Motor Score at Week 24 Using LOCF
Description: The UPDRS, a clinician-based rating scale, assesses 6 features of PD impairment: (1) mentation, behavior, and mood; (2) activities of daily living; (3) motor examination; (4) complications of therapy; (5) modified Hoehn and Yahr stage; (6) Schwab and England activities of daily living scale. Assessments were conducted when participants had benefit in regard to mobility, tremor, and rigidity. The total motor score (sum of motor examination) ranges from 0 to 108: 0=normal/no symptoms; 108=worst possible case. Change from BL was calculated as the value at Week 24 minus the value at BL.
Time Frame: Baseline and Week 24 (Visit 13)
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed. Data were collected using the LOCF method.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ropinirole PR
Number analyzed (Participants) | 167 | 174
scores on a scale | -0.7 (9.03) | -6.3 (10.08)

3. Secondary Outcome: Mean Change From Baseline in the Percentage of Awake Time Spent "Off" (ATSO) at Week 24 Using LOCF
Description: The "off" state is defined as the state in which PD symptoms (lack of mobility, tremor, or rigidity) are not adequately controlled by the drug. Participants were asked to record the duration of their "off" periods in 24-hour diary cards prior to each visit on the same 2 days of each relevant week. The total number of awake hours spent "off" per 24-hour period was the sum of the hours recorded on the two 24-hour diary cards. The percentage of ATSO=ATSO divided by (ATSO + awake time spent "on") * 100. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline.
Time Frame: Baseline and Week 24
Population: ITT Population. Data were collected using the LOCF method.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Placebo | Ropinirole PR
Number analyzed (Participants) | 169 | 175
Percentage of time | -1.8 (15.88) | -13.5 (15.62)

4. Secondary Outcome: Mean Change From Baseline in Total Awake Time Spent "on" at Week 24 Using LOCF
Description: The "on" state is defined as the state in which the PD symptoms (lack of mobility, tremor, or rigidity) are adequately controlled by the drug. Participants were asked to record the duration of their "on" periods in 24-hour diary cards prior to each visit on the same two days of each relevant week. The total number of awake hours spent "on" per 24-hour period was the sum of the hours recorded on the two 24-hour diary cards. Change from Baseline is calculated as the value at Week 24 minus the Baseline value.
Time Frame: Baseline and Week 24
Population: ITT Population. Data were collected using the LOCF method.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | Ropinirole PR
Number analyzed (Participants) | 169 | 175
hours | 0.1 (2.48) | 1.9 (2.44)

5. Secondary Outcome: Mean Change From Baseline in Total Awake Time "on" Without Troublesome Dyskinesias (TD) at Week 24 Using LOCF
Description: Dyskinesias are involuntary twisting, turning movements caused by medication during "on" time in PD. TD is defined as those movements that interfere with function and cause meaningful discomfort. Participants were asked to record the number of awake hours spent "on" without TD in 24-hour diary cards prior to each visit on the same two days of each relevant week. The total number of awake hours spent"on"without TD per 24-hour period was the sum of the hours recorded on the two 24-hour diary cards. Change from Baseline is calculated as the value at Week 24 minus the Baseline value.
Time Frame: Baseline and Week 24
Population: ITT Population. Data were collected using the LOCF method.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | Ropinirole PR
Number analyzed (Participants) | 169 | 175
hours | 0.3 (2.56) | 1.7 (2.81)

6. Secondary Outcome: Mean Change From Baseline in the UPDRS Activities of Daily Living (ADL) Score at Week 24 Using LOCF
Description: The UPDRS assesses six features of PD impairment, including Activities of Daily Living (ADL). The total ADL score ranges from 0 to 52, where 0= normal/no symptoms and 52= worst possible case. Change from Baseline is calculated as the value at Week 24 minus the Baseline value.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ropinirole PR
Number analyzed (Participants) | 167 | 174
scores on a scale | -0.2 (3.64) | -2.2 (3.93)

7. Secondary Outcome: Number of Responders Based on the Clinical Global Impression (CGI) Global Improvement Scale Using LOCF
Description: The CGI global improvement scale allows the investigator to rate the participant's total improvement since the beginning of treatment (Baseline). Scores on the scale range from 1 to 7 (1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse). Participants with a CGI global improvement score of <=2 (representing much improved or very much improved) were considered to be responders.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Ropinirole PR
Number analyzed (Participants) | 168 | 174
participants | 16 | 77

8. Secondary Outcome: Number of Participants Requiring Reinstatement of L-dopa Following a Dose Reduction Using LOCF
Description: In the event of unacceptable side effects relative to Baseline (e.g., dyskinesias, dystonias [neurological movement disorder]) the dosage of L-dopa was reduced. If there was reduction in the side effects and there was loss of symptom control, the dose of study medication was again increased (reinstated) at subsequent visits. If symptoms could still not be controlled, then L-dopa was reinstated; however, the dose could not exceed the baseline dose.
Time Frame: Week 24
Population: ITT Population. Only those participants who had their dose of L-dopa reduced were included in this analysis. Data were collected using the LOCF method.
Measure: Number; unit: participants
Arm/Group | Placebo | Ropinirole PR
Number analyzed (Participants) | 64 | 111
participants | 23 | 13

9. Secondary Outcome: Number of Responders to Study Treatment Using LOCF
Description: The "off" state is defined as the state in which PD symptoms (lack of mobility, tremor, or rigidity) are not adequately controlled by the drug. Responders are defined as participants who had at least a 20% reduction from Baseline in awake time spent "off" and at least a 20% reduction from Baseline in the L-dopa dose.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Ropinirole PR
Number analyzed (Participants) | 162 | 171
participants | 4 | 39

10. Secondary Outcome: Mean Change From Baseline in the Depression Scores on the Hamilton Depression Rating Scale (HAMD-17) Using LOCF
Description: The HAMD-17 is a 17-item scale that is completed by the investigator. Each item was evaluated and scored using either a 5-point scale (e.g., absent, mild, moderate, severe, very severe) or a 3-point scale (e.g., absent, mild, marked). The total HAMD-17 score (sum of the scores of all 17 items) may range from 0 (least severe) to 52 (most severe). Change from Baseline is calculated as the value at Week 24 minus the Baseline value.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ropinirole PR
Number analyzed (Participants) | 161 | 170
scores on a scale | -0.6 (4.33) | -1.6 (4.38)

11. Secondary Outcome: Mean Change From Baseline (BL) in the Parkinson's Disease Sleep Scale (PDSS) Total Score Using LOCF
Description: The PDSS uses a series of 15 questions to assess sleep disturbance associated with PD. Participants completed the assessments based on their experiences in the past week by marking a cross on each 10 centimeter (cm) scale (labelled from worst to best state). Responses were quantified by measuring the distance along each line where the cross was placed. The scores for each item ranged from 0 (symptom severe and always experienced) to 10 (symptom free). The maximum cumulative score for the PDSS was thus 150 (free of all symptoms). Change from BL=value at Week 24 minus the BL value.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ropinirole PR
Number analyzed (Participants) | 159 | 170
scores on a scale | -1.7 (20.57) | 0.5 (21.22)

12. Secondary Outcome: Mean Change From Baseline in the Parkinson's Disease Quality of Life Scores (PDQ39) Using LOCF
Description: The PDQ39 is a 39 item self-administered questionnaire. The questionnaire covers eight domains of health that are reported as adversely affected by patients with PD. Participants were asked to rate responses on a scale from 0 to 4 ("never" to "always"). The overall index score is the mean of the eight individual domain scores measured on a continuous scale ranging from 0 (no problem at all) to 100 (maximum level of the problem). Change from Baseline is calculated as the value at Week 24 minus the Baseline value.
Time Frame: Baseline and Week 24
Population: ITT Population. Only those participants contributing data at the indicated time points for the indicated domain were analyzed. Data were collected using the LOCF method.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ropinirole PR
Number analyzed (Participants) | 160 | 170
scores on a scale
  Mobility Domain; n=160, 170 | 2.5 (17.30) | -5.7 (18.10)
  Activities of Daily Living Domain; n=160, 170 | -0.3 (18.65) | -5.9 (18.20)
  Emotional Wellbeing Domain; n=160, 170 | -0.8 (15.30) | -4.8 (17.37)
  Stigma Domain; n=160, 170 | -1.1 (18.17) | -5.1 (18.01)
  Social Support Domain; n=157, 167 | -0.7 (15.21) | -0.4 (14.63)
  Cognitive Impairment Domain; n=160, 170 | -0.8 (13.28) | -1.1 (14.36)
  Communication Domain; n=160, 170 | 2.6 (17.21) | -1.1 (12.28)
  Bodily Discomfort Domain; n=160, 170 | 0.7 (19.15) | -3.5 (19.16)

13. Secondary Outcome: Time to Reinstatement of L-dopa Following a Reduction in Dose Using LOCF
Description: The mean number of days after which the dose of L-dopa was readministered after the reduction in dose was recorded.
Time Frame: Baseline to Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Ropinirole PR
Number analyzed (Participants) | 64 | 111
days | 114.3 (4.69) | 162.9 (3.55)

ADVERSE EVENTS:
Time Frame: Adverse event (AE) and serious adverse event (SAE) data are presented for the On-treatment Phase (Week 1 to Week 24) plus the 7-day Down-titration Period.
Description: SAEs and non-serious AEs were collected in the Safety Population, consisting of all participants who received at least one dose of randomized study medication (placebo or active drug). This does not include placebo given during the Placebo Run-in Period.
Arm/Group | Placebo | Ropinirole PR
Serious Adverse Events (participants affected / at risk) | 8/170 | 9/175
Other Adverse Events (participants affected / at risk) | 105/170 | 129/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=170) | Ropinirole PR (N=175)
Coronary artery disease (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Hernia (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Akinesia (Nervous system disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=170) | Ropinirole PR (N=175)
Dyskinesia (Nervous system disorders) | 5 | 31
Dizziness (Nervous system disorders) | 12 | 16
Somnolence (Nervous system disorders) | 7 | 10
Headache (Nervous system disorders) | 3 | 3
Akinesia (Nervous system disorders) | 3 | 2
Hypoaesthesia (Nervous system disorders) | 3 | 1
Parkinson's disease (Nervous system disorders) | 2 | 2
Sciatica (Nervous system disorders) | 0 | 3
Dyspraxia (Nervous system disorders) | 0 | 2
Lethargy (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 1 | 1
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dystonia (Nervous system disorders) | 0 | 1
Head titubation (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Narcolepsy (Nervous system disorders) | 1 | 0
Parkinsonian gait (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Vascular headache (Nervous system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 10 | 10
Nausea (Gastrointestinal disorders) | 5 | 10
Diarrhea (Gastrointestinal disorders) | 4 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 3
Abdominal discomfort (Gastrointestinal disorders) | 1 | 4
Toothache (Gastrointestinal disorders) | 0 | 4
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 2 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 6 | 4
Edema peripheral (General disorders) | 4 | 5
Fatigue (General disorders) | 2 | 6
Chest discomfort (General disorders) | 2 | 0
Disease progression (General disorders) | 1 | 1
Gait disturbance (General disorders) | 1 | 1
Hernia (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Discomfort (General disorders) | 1 | 0
Face edema (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Swelling (General disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 6 | 6
Hallucination (Psychiatric disorders) | 4 | 7
Sleep disorder (Psychiatric disorders) | 1 | 2
Abnormal dreams (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Illusion (Psychiatric disorders) | 0 | 2
Nightmare (Psychiatric disorders) | 0 | 2
Dependence (Psychiatric disorders) | 1 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0
Hypersexuality (Psychiatric disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 7 | 6
Hypertension (Vascular disorders) | 6 | 1
Hypotension (Vascular disorders) | 1 | 4
Angiopathy (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0
Orthostatic hypertension (Vascular disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 6
Pneumonia (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1
Impetigo (Immune system disorders) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 11 | 12
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Palpitations (Cardiac disorders) | 6 | 4
Arrhythmia (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 1 | 1
Cardiac discomfort (Cardiac disorders) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Weight decreased (Investigations) | 6 | 2
Blood pressure increased (Investigations) | 3 | 4
Blood pressure decreased (Investigations) | 1 | 0
Neutrophil count abnormal (Investigations) | 0 | 1
Vision blurred (Eye disorders) | 4 | 3
Cataract (Eye disorders) | 1 | 1
Conjunctival hyperemia (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Exophthalmos (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Night blindness (Eye disorders) | 1 | 0
Oculogyric crisis (Eye disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 2
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 6
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 2
Chromaturia (Renal and urinary disorders) | 0 | 1
Incontinence (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Spermatorrhea (Reproductive system and breast disorders) | 0 | 1
Gambling (Social circumstances) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.